CLINICAL TRIAL: NCT04703036
Title: Randomized Trial of Supplementing Glycine and N-acetylcysteine vs. Placebo in COVID-19
Brief Title: Glutathione, Oxidative Stress and Mitochondrial Function in COVID-19
Status: Terminated | Phase: Early Phase 1 | Type: Interventional
Why Stopped: Futility due to inability to recruit participants meeting entry criteria.
Sponsor: Baylor College of Medicine (Other)
Responsible Party: Principal Investigator, Rajagopal V Sekhar, Principal Investigator, Baylor College of Medicine
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: H48057
Record Dates: First submitted 2021-01-06; First posted 2021-01-11 (Actual); Last update posted 2024-06-26 (Actual); Status verified 2024-06

CONDITIONS: Covid19
MeSH Terms: conditions — COVID-19 | interventions — Glycine; Acetylcysteine; Alanine

STUDY DESIGN:
Intervention Model Description: Randomized controlled trial, placebo-controlled, double-blind design
Who Masked: Participant, Investigator
Masking Description: Participants and the investigative team are masked. Only the biostatistician will be unmasked to the identity of the active and placebo groups.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active arm (Experimental): The active supplements are glycine and N-acetylcysteine
  Interventions: Dietary Supplement: Glycine; Dietary Supplement: N-acetylcysteine
- Placebo arm (Placebo Comparator): The placebo arm is alanine
  Interventions: Dietary Supplement: Alanine

INTERVENTIONS:
Dietary Supplement: Glycine — Glycine is an amino-acid (protein)
  Arms: Active arm
Dietary Supplement: N-acetylcysteine — This is a donor of the amino-acid cysteine (protein)
  Arms: Active arm
Dietary Supplement: Alanine — Alanine is an amino-acid (protein)
  Arms: Placebo arm

SUMMARY:
COVID-19 is associated with increased mortality, and has been linked to a 'cytokine inflammatory storm'. Populations at higher risk of COVID complications and mortality include the elderly, diabetic patients and immunocompromised patients (such as HIV), and the investigators have studied these 3 populations over the past 20 years and have found that they all have deficiency of the endogenous antioxidant protein glutathione (GSH), elevated oxidative stress, inflammation, impaired mitochondrial function, immune dysfunction, and endothelial dysfunction.

It is known and established that GSH adequacy is necessary for neutralizing harmful oxidative stress, and that elevated oxidative stress appears to promote mitochondrial dysfunction. The combination of oxidative stress and mitochondrial dysfunction have also been linked to inflammation, immune dysfunction, and endothelial dysfunction. In prior studies in aging, the investigators have also identified that supplementing glutathione precursor amino-acids glycine and cysteine (provided as N-acetylcysteine) improves GSH deficiency and mitochondrial function, and lowers oxidative stress, inflammation, and endothelial dysfunction. The investigators have coined the term GlyNAC to refer to the combination of glycine and N-acetylcysteine.

This study will evaluate the prevalence and extent of these defects in patients with COVID-19 admitted to the hospital, and the response to supplementing GlyNAC or placebo for 2-weeks. Because patients with COVID-19 are also being reported to have fatigue and cognitive impairment, the investigators will also measure fatigue and cognition at admission, 1-week and 2-weeks after beginning supplementation. The supplementation is stopped after completing 2-weeks, and these outcomes will be measured again after 4-weeks and 8-weeks after stopping supplementation.

DETAILED DESCRIPTION:
This study will investigate associated defects in the following two populations of patients with COVID-19:

Hospitalized patients admitted for COVID-19 will sign an informed consent form, and be randomized to receive either active (Glycine plus N-acetylcysteine) or a placebo (alanine) supplementation for 2-weeks. On day-0, the participants will have a single blood draw to measure measure oxidative stress, Glutathione levels, inflammatory cytokines, endothelial dysfunction, mitochondrial dysfunction, immune dysfunction, and complete questionnaires to assess fatigue, activity and cognition. Additional clinical and lab information will be obtained from the hospital electronic medical records. These measurements will be repeated 1-week and 2-weeks after starting supplementation, and at 4-weeks and 8-weeks after stopping supplementation.

ELIGIBILITY:
Inclusion Criteria:

* Age 55-85y;
* Diagnosis of COVID-19;
* Hospitalized patients.

Exclusion Criteria:

* Active heart disease or active cancer at time of recruitment;
* Patients in Intensive Care Unit at the time of recruitment;
* Patents with alanine transaminase and aspartate transaminase greater than 5 times the upper limit of normal at any time;
* Patients requiring >4L per minute of oxygen support at the time of recruitment.

Ages: 55 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2021-01-11 (Actual); Primary Completion 2023-03-31 (Actual); Study Completion 2023-03-31 (Actual)

PRIMARY OUTCOMES:
Change in Glutathione concentrations | Day 0, 3-days, 1-week, 2-weeks, 6-weeks, 10-weeks
  Glutathione levels will be measured in red-blood cells
Change in Interleukein 6 concentrations | Day 0, 3-days, 1-week, 2-weeks, 6-weeks, 10-weeks
  Plasma IL-6 concentrations
Change in Ordinal scale | Day 0, 1-week, 2-weeks
  This is a scale developed by the World-Health Organization for COVID trials. The clinical condition of each participant will be determined using this scale at 3 time points - Day 0, after 1-week and after-2weeks of supplementation

SECONDARY OUTCOMES:
Change in oxidative stress | Day 0, 1-week, 2-weeks, 6-weeks, 10-weeks
  Plasma concentrations of TBARS
Change in marker of damage due to oxidative stress | Day 0, 1-week, 2-weeks, 6-weeks, 10-weeks
  Plasma concentrations of F2-isoprostanes
Change in inflammatory cytokines | Day 0, 1-week, 2-weeks, 6-weeks, 10-weeks
  Plasma concentrations of TNFa, hsCRP, IL-10, PAI-1, D-dimer
Change in mitochondrial energetics | Day 0 1-week, 2-weeks, 6-weeks, 10-weeks
  Energetics measured by high-resolution respirometry in peripheral blood monocytes
Change in immune function | Day 0, 1-week, 2-weeks, 6-weeks, 10-weeks
  The trial will evaluate if COVID-related disease severity is associated with NK cell deficiency and antigen presenting cell production of IL-6 and TNF.
Change in cognition | Day 0, 1-week, 2-weeks, 6-weeks, 10-weeks
  Measured using Montreal cognitive assessment which ranges from 0-30
Change in function | Day 0, 1-week, 2-weeks, 6-weeks, 10-weeks
  Measured using the Katz-activities of daily living
Change in fatigue | Day 0, 1-week, 2-weeks, 6-weeks, 10-weeks
  Measured using the Facit-F fatigue scale
Change in circulating marker of memory | Day 0, 1-week, 2-weeks, 6-weeks, 10-weeks
  Plasma BDNF concentrations

CONTACTS AND LOCATIONS:
Locations (1):
- Baylor College of Medicine, Houston, Texas, United States